CLINICAL TRIAL: NCT04989569
Title: Serial Body Composition Change for Risk Prediction and Nutritional Guide in Treating Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201901875A3C501
Record Dates: First submitted 2021-07-01; First posted 2021-08-04 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Sepsis
Keywords: sepsis; body composition; Nutritional intervention
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The investigators will use the random number generator to divide the patients into two groups, the control group (with no nutritional intervention) and the intervention group (with nutritional intervention). The body composition data (of day 1, 3, 8) of the patients in the control group will not be given to the dietitians for adjusting the diet formula according to the patient's body composition.
- nutritional intervention (Experimental): The investigators will use the random number generator to divide the patients into two groups, the control group (with no nutritional intervention) and the intervention group (with nutritional intervention). The body composition data (of day 1, 3, 8) of the patients in the intervention group will be given to the dietitians for adjusting the diet formula according to the patient's body composition.
  Interventions: Dietary Supplement: Nutritional intervention

INTERVENTIONS:
Dietary Supplement: Nutritional intervention — In the intervention group, the body composition data (of day 1, 3, 8) will be given to the dietitians for adjusting the diet formula. The diet formula will be adjusted on the discretion of the dietitian caring for the septic patients based on clinical judgement. The policy adopted by the dietary treatment guidelines for sepsis is to adjust the dietary concentration when there is too much extracellular water under the premise of gastrointestinal tolerance. When the skeletal muscle mass loss is too fast, the dietitians will increase the protein intake by 1.2g/kg of body weight. For patients with acute renal failure and excess extracellular water accumulation and muscle loss, the dietitians will adjust the protein, sodium, potassium, calcium and phosphorus content in the formula. The dietitians will give appropriate nutrition prescriptions based on clinical signs, disease diagnosis and biochemical values.
  Arms: nutritional intervention

SUMMARY:
To explore whether serial changes of data in body composition of patients with sepsis can help clinician to monitor prognosis.

DETAILED DESCRIPTION:
The investigators will use the random number generator to divide the patients into two groups, the control group (with no nutritional intervention) and the intervention group (with nutritional intervention). The body composition data (of day 1, 3, 8) of the patients in the intervention group will be given to the dietitians for adjusting the diet formula according to the patient's body composition.The patients in control group also will undergo Bio-electrical Impedance Analysis (BIA) assessment, but not disclosed to the dietitian. The diet formula will be adjusted on the discretion of the dietitian caring for the septic patients based on clinical judgement.

ELIGIBILITY:
Inclusion Criteria:

1. ICU patient
2. Clinical diagnosis of sepsis

Exclusion Criteria:

1. Expired within 3-days

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
ICU mortality | The day discharged from ICU, an average of 2 weeks
  Status of survival or mortality at the time discharged from ICU
Hospital mortality | The day discharged from hospital, an average of 5 weeks
  Status of survival or mortality at the time discharged from hospital
7-day mortality | Day 7 after hospital admission
  Status of survival or mortality at Day 7 during hospital stay
28-day mortality | Day 28 after hospital admission
  Status of survival or mortality at Day 28 during hospital stay
90-day mortality | Day 90 after hospital admission
  Status of survival or mortality at Day 90 during hospital stay

SECONDARY OUTCOMES:
Change of white blood cell between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of white blood cell count between day 1 and day 3
Change of white blood cell between day 1 and day 8 | Day 1 and Day8 after ICU admission
  assessing the change of white blood cell count between day 1 and day 8
Change of white blood cell between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of white blood cell count between day 3 and day 8
Change of pulse pressure between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of pulse pressure between day 1 and day 3
Change of pulse pressure between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of pulse pressure between day 1 and day 8
Change of pulse pressure between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of pulse pressure between day 3 and day 8
Day 1 Sequential Organ Failure Assessment score | Day 1 after ICU admission
  assessing Sequential Organ Failure Assessment score at day 1
Day 3 Sequential Organ Failure Assessment score | Day 3 after ICU admission
  assessing Sequential Organ Failure Assessment score at day 3
Day 8 Sequential Organ Failure Assessment score | Day 8 after ICU admission
  assessing Sequential Organ Failure Assessment score at day 8
Ventilation days | The day weaned off ventilator, an average of 3 weeks
  Total using days of mechanical ventilation
Change of percentage of body fat between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of percentage of body fat between day 1 and day 3
Change of percentage of body fat between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of percentage of body fat between day 1 and day 8
Change of percentage of body fat between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of percentage of body fat between day 3 and day 8
Change of protein intake between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of protein intake (g/day, g/kg) between day 1 and day 3
Change of protein intake between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of protein intake (g/day, g/kg) between day 1 and day 8
Change of protein intake between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of protein intake (g/day, g/kg) between day 3 and day 8
Change of energy intake between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of energy intake (total kcal/day) between day 1 and day 3
Change of energy intake between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of energy intake (total kcal/day) between day 1 and day 8
Change of energy intake between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of energy intake (total kcal/day) between day 3 and day 8
Change of segment/monocyte ratio between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of segment count to monocyte count ratio between day 1 and day 3
Change of segment/monocyte ratio between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of segment count to monocyte count ratio between day 1 and day 8
Change of segment/monocyte ratio between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of segment count to monocyte count ratio between day 3 and day 8
Change of total body water between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of total body water between day 1 and day 3
Change of total body water between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of total body water between day 1 and day 8
Change of total body water between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of total body water between day 3 and day 8
Change of soft lean mass between day 1 and day 3 | Day 1 and Day 3 after ICU admission
  assessing the change of soft lean mass between day 1 and day 3
Change of soft lean mass between day 1 and day 8 | Day 1 and Day 8 after ICU admission
  assessing the change of soft lean mass between day 1 and day 8
Change of soft lean mass between day 3 and day 8 | Day 3 and Day 8 after ICU admission
  assessing the change of soft lean mass between day 3 and day 8
ICU Days | The day discharged from ICU, an average of 2 weeks
  length of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: FANG WEN-FENG, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan